CLINICAL TRIAL: NCT04960995
Title: Description of Case of Infection With a New Species of Babesia and Its Molecular Diagnosis
Acronym: BADIAG
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8341
Record Dates: First submitted 2021-07-02; First posted 2021-07-14 (Actual); Last update posted 2021-07-23 (Actual); Status verified 2021-07

CONDITIONS: Babesiosis, Human
Keywords: Babesiosis; BABESIA; ZOONOSES
MeSH Terms: conditions — Babesiosis; Zoonoses

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Babesiosis is a potentially very serious infection, but too little known. investigators want to raise their clinical colleagues and remind fellow biologists of the importance of choosing a good molecular diagnosis so as not to give false-negative results.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Splenectomized subject
* Subject with severe babesiosis
* Subject not having expressed, after information, his opposition to the reuse of his data for the purposes of this research

Exclusion criteria:

- Subject having expressed opposition to participating in the study

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject suffering from severe babesiosis
Sampling Method: Non-Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2021-07-10 (Actual); Primary Completion 2021-07-15 (Estimated); Study Completion 2021-07-15 (Estimated)

PRIMARY OUTCOMES:
A retrospective study describing a case of infection with a new species of Babesia | The files analyzed retrospectively concern the period from January 01, 2020 to December 31, 2020.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander PFAFF, MCU-PH, Principal Investigator — Parasitology and Medical Mycology Department - Strasbourg University Hospitals
Locations (1):
- Parasitology and Medical Mycology Department - Strasbourg University Hospitals, Strasbourg, France